CLINICAL TRIAL: NCT07063225
Title: Romiplostim N01 for Chemotherapy-induced Thrombocytopenia in Tumors: a Prospective Multi-center One-arm Study
Brief Title: Romiplostim N01 for Chemotherapy-induced Thrombocytopenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other); Tianjin Medical University Second Hospital (Other); Tianjin Third Central Hospital (Other); Tianjin People's Hospital (Other); Henan Cancer Hospital (Other Government); The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025061
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-06

CONDITIONS: Chemotherapy-induced Thrombocytopenia; Romiplostim N01

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Romiplostim N01 (Experimental): 50 enrolled subjects will be picked up to take Romiplostim N01 at the indicated dose.
  Interventions: Drug: Romiplostim N01

INTERVENTIONS:
Drug: Romiplostim N01 — The subjects will receive ropivacaine N01 treatment, with an initial dose of (2-3) µg/kg. When the dose is less than 250 µg, 250 µg (1 vial) can be administered (subcutaneously), once a week. The dose will be increased by (1) µg/kg each week, up to a maximum of 10 µg/kg, until the platelet count reaches ≥ 50 × 10^9/L. If the platelet count returns to normal, the dose can be reduced according to the platelet level as appropriate.

SUMMARY:
To evaluate the efficacy and safety of Romiplostim N01 to treat chemotherapy-induced thrombocytopenia in tumors

DETAILED DESCRIPTION:
The investigator had registered a clinical trial of Eltrombopag in the treatment of chemotherapy-induced thrombocytopenia（NCT04600960）. Due to the late launch of Romiplostim N01 in China, the investigator also collected the information of Romiplostim N01 in the treatment of chemotherapy-induced thrombocytopenia according to the protocal of Eltrombopag in the treatment of chemotherapy-induced thrombocytopenia（NCT04600960）.

This is a single-arm study to evaluate the safety and efficacy of Romiplostim N01 to treat chemotherapy-induced thrombocytopenia （CIT）in tumors. These subjects have been treated with recombinant human thrombopoietin（rhTPO） or interleukin 11（IL-11） before, the platelets can rise to normal or reach the effective standard, but after the re-application, the effective standard is not reached, or the effective standard is still not reached after the rhTPO 300U/kg/d treatment for 14 days. The investigator will assess the changes of the platelet counts after the treatment of Romiplostim N01 from week 1 to week 24, and observe incidence of adverse events during the treatment of Romiplostim N01. The investigator will complete the 4 weeks safety visits（once a week），if the subjects end or withdraw from the clinical trial.

Patients with chemotherapy-induced thrombocytopenia who had the same inclusion and exclusion criteria in the same period or in the past will be compared with the efficacy and safety of supportive treatment and Eltrombopag in the same period or history, so as to preliminarily explore and evaluate the efficacy and safety of Romiplostim N01 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years or above, gender not restricted;
* Patients who meet the diagnostic criteria for chemotherapy-related thrombocytopenia, and still ineffective after repeated treatment with rhTPO or IL-11 (subjects need to undergo regular rhTPO treatment for at least 14 days after radiotherapy and chemotherapy, with a dose of rhTPO 300u/kg/d or higher, and the platelet count remains less than 30×10^9/L, defined as refractory CTIT);
* Patients who have stopped chemotherapy and radiotherapy for more than 1 month;
* Patients with platelet count at enrollment < 30×10^9/L;
* Patients with platelet count remains < 30×10^9/L for more than 1 month;
* Patients with expected survival period ≥ 6 months;
* Patients with liver and kidney function < 1.5× upper limit of normal value, physical examination qualified;
* Patients with ECOG physical status score ≤ 2 points;
* Patients with Cardiac function: New York Heart Association cardiac function classification is grade 2 or below;
* Patients who is voluntary to sign the informed consent form;

Exclusion Criteria:

* Those with uncontrollable primary diseases of important organs, such as extensive metastasis of malignant tumors, liver failure, heart failure, kidney failure and other diseases；
* Patients with poor compliance;
* Positive serology for HIV, hepatitis B virus (HBV), hepatitis C virus (HCV), and/or hepatitis D virus (HDV), Syphilis; Positive for Epstein-Barr Virus DNA, Cytomegalovirus DNA;
* Accompanied by extensive and severe bleeding, such as hemoptysis, upper gastrointestinal bleeding, intracranial hemorrhage, etc.
* There is currently a heart disease requiring treatment or a poorly controlled hypertension judged by the investigator；
* Patients with thrombotic diseases such as pulmonary embolism, thrombosis, and atherosclerosis；
* Those who have received allogeneic stem cell transplantation or organ transplantation in the past；
* Patients with mental disorders who cannot normally obtain informed consent and undergo trials and follow-up；
* Patients whose toxic symptoms caused by treatment before participating in the trial have not disappeared；
* Other serious diseases that may restrict participants from participating in this trial (such as diabetes; severe heart failure; myocardial obstruction or unstable arrhythmia or unstable angina in the past 6 months; gastric ulcers; mobility Autoimmune diseases, etc.)；
* Patients with sepsis or patients with other irregular bleeding；
* Patients taking antiplatelet drugs at the same time；
* Pregnant women, suspected pregnancy (a positive pregnancy test for human chorionic gonadotropin in urine at screening) and breastfeeding patients； Pre-existing cardiac disease, including congestive heart failure of New York Heart Association [NYHA] Grade III/IV, arrhythmia requiring treatment or myocardial infarction within the last 6 months. No arrhythmia known to increase the risk of thrombotic events (e.g. atrial fibrillation), or patients with a QT >450msec or QTc > 480 for patients with a Bundle Branch Block;
* Researchers believe that patients should not participate in the test of any other condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Efficiency after 12 weeks of treatment with Romiplostim N01 | 12 weeks
  The proportion of patients whose platelet count was ≥ 50 × 10^9/L after 12 weeks (3 months) of treatment with Romiplostim N01.

SECONDARY OUTCOMES:
Other efficacy evaluation after 12 weeks of treatment with Romiplostim N01 | 12 weeks
  The proportion of patients whose platelet count was ≥ 30×10^9/L or ≥ 100×10^9/L after 12 weeks (3 months) of treatment with Romiplostim N01
Efficiency after 24 weeks of treatment with Romiplostim N01 | 24 weeks
  The proportion of patients whose platelet count was ≥ 30×10^9/L, ≥ 50×10^9/L, or ≥ 100×10^9/L after 24 weeks (6 months) of treatment with Romiplostim N01
Platelet counts at each visit point | 24 weeks
  Platelet counts after the treatment of Romiplostim N01 at each visit point
WHO bleeding scale at each visit point | 24 weeks
  Changes of the WHO bleeding scale after the treatment of Romiplostim N01 at each visit point. The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Adverse events | 24 weeks
  Incidence, severity, and relationship of treatment emergent adverse events after Romiplostim N01 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yunfei Chen, MD, Principal Investigator — Chinese Academy of Medical Science and Blood Disease Hospital
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months to 36 months after study completion.
Supporting Information: SAP, ICF
Time Frame: 12 months to 36 months after study completion.
Access Criteria: Upon request to PI.